CLINICAL TRIAL: NCT01836861
Title: A Phase 1, Open-Label Study of the Absorption, Distribution, Metabolism and Excretion of 14C-Labeled IPI-145 and the Absolute Bioavailability of IPI-145 in Healthy Subjects
Brief Title: IPI-145 ADME and Absolute Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IPI-145-05; 2012-005425-75 (EudraCT Number)
Record Dates: First submitted 2013-04-01; First posted 2013-04-22 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Healthy
Keywords: Phase I; healthy male volunteers; ADME; Bioavailability; PI3K inhibitor; Absorption; Distribution; Metabolism; Excretion; safety
MeSH Terms: interventions — duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPI-145 and [14C] IPI-145 (Experimental)
  Interventions: Drug: IPI-145

INTERVENTIONS:
Drug: IPI-145 — Intravenous infusion: approximately 2.8 μg IPI-145 containing 14.8 kBq of radioactivity; Oral suspension: 25 mg IPI-145 containing approximately 3.15 MBq of radioactivity; Oral capsule: 25 mg IPI-145

SUMMARY:
This is an open-label, 2-period, absorption, distribution, metabolism and excretion (ADME) and absolute bioavailability study in 6 healthy adult male subjects.

DETAILED DESCRIPTION:
In Period 1, subjects will receive a single oral dose of 25 mg IPI-145, followed by a 15-minute IV infusion of approximately 2.8 μg 14C-IPI-145 containing 14.8 kBq of radioactivity.

In Period 2, the same subjects will receive a single dose of 25 mg 14C-IPI-145 as an oral suspension, containing approximately 3.15 MBq of radioactivity.

There will be a washout period of at least 14 days between Period 1 and Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Males, between 18 and 45 years of age, inclusive Body Mass Index (BMI) : 18.0-30.0 kg/m2
* In good health, determined by no clinically significant findings from medical history, physical examination (Check-in), 12-lead ECG, and vital signs
* Provision of signed and dated, written informed consent prior to any study specific procedures

Exclusion Criteria:

* Evidence of clinically significant medical conditions
* History of gastrointestinal surgery that may affect drug absorption
* Positive or indeterminate QuantiFERON-TB Gold test at screening
* Any active infection at the time of screening or admission
* Participation in another ADME study with a radiation burden >0.1 mSv in the period of 1 year before screening
* Irregular defecation pattern (less than once per 2 days)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-03; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
PK parameters (AUC) of IPI-145 in plasma | over 48 hours
PK parameters (AUC) and radioactivity excreted in urine and feces | over 144 hours
PK parameters (Cmax) of IPI-145 in plasma | over 48 hours
PK parameters (t1/2) of IPI-145 in plasma | over 48 hours
PK parameters (Cmax) and radioactivity excreted in urine and feces | over 144 hours
PK parameters (t1/2) and radioactivity excreted in urine and feces | over 144 hours

SECONDARY OUTCOMES:
Number of participants with adverse events following a single dose administration of IPI-145 | over 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (1):
- Pharmaceuticals Research Association (PRA), Zuidlaren, Netherlands